CLINICAL TRIAL: NCT05648110
Title: A Phase I/III Randomized, Double-blind Study to Evaluate the Safety, Efficacy and Neutralizing Activity of AZD5156/AZD3152 for Pre-exposure Prophylaxis of COVID-19 in Participants With Conditions Causing Immune Impairment. Sub-study: Phase II Open Label Sub-study to Evaluate the Safety, PK, and Neutralizing Activity of AZD3152 for Pre-exposure Prophylaxis of COVID-19
Brief Title: Study Understanding Pre-Exposure pRophylaxis of NOVel Antibodies (SUPERNOVA) Sub-study: Study Understanding Pre-Exposure pRophylaxis of NOVel Antibodies (SUPERNOVA) Sub-study
Acronym: SUPERNOVA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D7000C00001; 2024-512554-15-00 (Registry Identifier: EU CT number); 2022-002378-95 (EudraCT Number)
Record Dates: First submitted 2022-11-30; First posted 2022-12-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: COVID-19, SARS-CoV-2
Keywords: Pre-exposure Prophylaxis of COVID-19
MeSH Terms: conditions — COVID-19 | interventions — cilgavimab and tixagevimab drug combination

STUDY DESIGN:
Intervention Model Description: D7000C00001 is a Phase I/III study (Parent study) being conducted in conjunction with a Phase II sub study that will be conducted in approximately 3706 participants (approximately 3256 in the Parent study and 450 in the sub study) to evaluate the safety, efficacy, PK, and neutralizing activity of AZD3152 compared with comparator for pre exposure prophylaxis of COVID-19, and separately evaluate the safety and PK of AZD5156, a combination of AZD3152 and AZD1061.
  The Parent study will consist of 2 cohorts: a Sentinel Safety Cohort and a Main Cohort. The Sentinel Safety Cohort will compare AZD5156 with placebo, while the Main Cohort will compare AZD3152 with placebo.
  The sub-study will have an initial Sentinel Safety Cohort that will include 12 healthy volunteers; all other participants in the study will be either immunocompromised or immunocompetent with all degrees of SARS-CoV-2 infection risk. Participants will be randomized 2:1 to receive AZD3152 or AZD7442 (EVUSHELD).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: For the Sentinel Safety Cohort and Main Cohort, neither the participant nor any of the Investigators or Sponsor staff who are involved in the treatment or clinical evaluation and monitoring of the participants will be aware of the study intervention received. Since AZD5156, AZD3152, and placebo are visually distinct prior to dose preparation (due to differences in vial volumes and container closure), study intervention will be handled by an unblinded pharmacist and administered by an unblinded administrator (or designee, in accordance with local and institutional regulations) at the study site who will be independent of safety evaluations and other trial evaluations. Personnel preparing and administering study intervention may be the same individual. Syringe masking will be required in order to maintain the blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Parent study Sentinel Safety Cohort - Subcohort 1a Gluteal - AZD5156 (Experimental): The Sentinel Safety Cohort of the Parent Study will enroll 56 healthy adults, 18 to 55 years of age, who will be randomized to receive AZD5156 (40 participants) or placebo (16 participants). Participants will be randomized to receive study intervention IM either in the gluteal or the anterolateral thigh. Dosing within the Sentinel Safety Cohort will be staggered, with participants allocated sequentially to 4 subcohorts (1a, 1b, 2a, and 2b).
  Interventions: Biological: AZD5156 (Parent study Sentinel Safety Cohort)
- Parent study Sentinel Safety Cohort - Subcohort 1a Gluteal - Placebo (Placebo Comparator): The Sentinel Safety Cohort of the Parent study will enroll 56 healthy adults, 18 to 55 years of age, who will be randomized to receive AZD5156 (40 participants) or placebo (16 participants). Participants will be randomized to receive study intervention IM either in the gluteal or the anterolateral thigh. Dosing within the Sentinel Safety Cohort will be staggered, with participants allocated sequentially to 4 subcohorts (1a, 1b, 2a, and 2b).
  Interventions: Biological: Placebo (Parent study Sentinel Safety Cohort)
- Parent study Sentinel Safety Cohort - Subcohort 1b Thigh - AZD5156 (Experimental): The Sentinel Safety Cohort of the Parent study will enroll 56 healthy adults, 18 to 55 years of age, who will be randomized to receive AZD5156 (40 participants) or placebo (16 participants). Participants will be randomized to receive study intervention IM either in the gluteal or the anterolateral thigh. Dosing within the Sentinel Safety Cohort will be staggered, with participants allocated sequentially to 4 subcohorts (1a, 1b, 2a, and 2b).
  Interventions: Biological: AZD5156 (Parent study Sentinel Safety Cohort)
- Parent study Sentinel Safety Cohort - Subcohort 1b Thigh - Placebo (Placebo Comparator): The Sentinel Safety Cohort of the Parent study will enroll 56 healthy adults, 18 to 55 years of age, who will be randomized to receive AZD5156 (40 participants) or placebo (16 participants). Participants will be randomized to receive study intervention IM either in the gluteal or the anterolateral thigh. Dosing within the Sentinel Safety Cohort will be staggered, with participants allocated sequentially to 4 subcohorts (1a, 1b, 2a, and 2b).
  Interventions: Biological: Placebo (Parent study Sentinel Safety Cohort)
- Parent study Sentinel Safety Cohort - Subcohort 2a Gluteal- AZD5156 (Experimental): The Sentinel Safety Cohort of the Parent study will enroll 56 healthy adults, 18 to 55 years of age, who will be randomized to receive AZD5156 (40 participants) or placebo (16 participants). Participants will be randomized to receive study intervention IM either in the gluteal or the anterolateral thigh. Dosing within the Sentinel Safety Cohort will be staggered, with participants allocated sequentially to 4 subcohorts (1a, 1b, 2a, and 2b).
  Interventions: Biological: AZD5156 (Parent study Sentinel Safety Cohort)
- Parent study Sentinel Safety Cohort - Subcohort 2a Gluteal - Placebo (Placebo Comparator): The Sentinel Safety Cohort of the Parent study will enroll 56 healthy adults, 18 to 55 years of age, who will be randomized to receive AZD5156 (40 participants) or placebo (16 participants). Participants will be randomized to receive study intervention IM either in the gluteal or the anterolateral thigh. Dosing within the Sentinel Safety Cohort will be staggered, with participants allocated sequentially to 4 subcohorts (1a, 1b, 2a, and 2b).
  Interventions: Biological: Placebo (Parent study Sentinel Safety Cohort)
- Parent study Sentinel Safety Cohort - Subcohort 2b Thigh - AZD5156 (Experimental): The Sentinel Safety Cohort of the Parent study will enroll 56 healthy adults, 18 to 55 years of age, who will be randomized to receive AZD5156 (40 participants) or placebo (16 participants). Participants will be randomized to receive study intervention IM either in the gluteal or the anterolateral thigh. Dosing within the Sentinel Safety Cohort will be staggered, with participants allocated sequentially to 4 subcohorts (1a, 1b, 2a, and 2b).
  Interventions: Biological: AZD5156 (Parent study Sentinel Safety Cohort)
- Parent study Sentinel Safety Cohort - Subcohort 2b Thigh - Placebo (Placebo Comparator): The Sentinel Safety Cohort of the Parent study will enroll 56 healthy adults, 18 to 55 years of age, who will be randomized to receive AZD5156 (40 participants) or placebo (16 participants). Participants will be randomized to receive study intervention IM either in the gluteal or the anterolateral thigh. Dosing within the Sentinel Safety Cohort will be staggered, with participants allocated sequentially to 4 subcohorts (1a, 1b, 2a, and 2b).
  Interventions: Biological: Placebo (Parent study Sentinel Safety Cohort)
- Parent study Main Cohort - AZD3152 (Experimental): The Main Cohort of the Parent study will enroll approximately 3200 participants. Dosing in the Main Cohort will be staggered, so that it starts with adult participants aged 18 years and older, with no adolescent participants dosed in the Main Cohort until safety data from Visit 2a (Day 8) and Visit 2b (Day 15) have been reviewed by the DSMB for at least 80 adult Main Cohort participants (which will include at least 40 participants who have received AZD3152). Participants in the Main Cohort will be randomized 1:1 to receive AZD3152 300 mg or comparator administered IM in the anterolateral thigh on Day 1. Participants will receive a second dose of their original randomized study intervention (ie, active treatment or comparator) 6 months after Visit 1.
  Interventions: Biological: Placebo (Parent study Sentinel Safety Cohort); Biological: AZD3152 (Parent study Main Cohort)
- Parent study Main Cohort - EVUSHELD™ (Active Comparator): Participants in the Main Cohort of the Parent study will be randomized 1:1 to receive AZD3152 300 mg or comparator administered IM in the anterolateral thigh on Day 1. Participants will receive a second dose of their original randomized study intervention (ie, active treatment or comparator) 6 months after Visit 1.
  At the request of regulatory authorities the active comparator will be changed to placebo. As the comparator is given on two occasions, this means that a participant randomized to the comparator arm may receive (a) two doses of EVUSHELD, (b) a dose of EVUSHELD and a dose of placebo, or (c) two doses of placebo.
  Interventions: Biological: EVUSHELD™ (Parent study Main Cohort)
- Parent study Main Cohort - Placebo (Placebo Comparator): Participants in the Main Cohort of the Parent study will be randomized 1:1 to receive AZD3152 300 mg or comparator administered IM in the anterolateral thigh on Day 1. Participants will receive a second dose of their original randomized study intervention (ie, active treatment or comparator) 6 months after Visit 1.
  At the request of regulatory authorities the active comparator will be changed to placebo. As the comparator is given on two occasions, this means that a participant randomized to the comparator arm may receive (a) two doses of EVUSHELD, (b) a dose of EVUSHELD and a dose of placebo, or (c) two doses of placebo.
  Interventions: Biological: Placebo (Parent study Main Cohort)
- Sub-study - AZD3152 (Experimental): This sub-study will enroll approximately 450 participants, ≥ 18 years of age with a minimum weight of 40 kg. An initial Sentinel Safety Cohort will include 12 healthy volunteers; all other participants in the study will be either immunocompromised or immunocompetent (including healthy participants) with all degrees of SARS-CoV-2 infection risk.
  Interventions: Biological: AZD3152 (Sub-study)
- Sub-study - AZD7442 (EVUSHELD™) (Active Comparator): This sub-study will enroll approximately 450 participants, ≥ 18 years of age with a minimum weight of 40 kg. An initial Sentinel Safety Cohort will include 12 healthy volunteers; all other participants in the study will be either immunocompromised or immunocompetent (including healthy participants) with all degrees of SARS-CoV-2 infection risk.
  Interventions: Biological: AZD7442 - EVUSHELD™ (Sub-study)
- Sub-study - AZD7442 (EVUSHELD™) Immunocompromised participants offered AZD3152 1200mg IV (Experimental): This sub-study will enroll approximately 450 participants, ≥ 18 years of age with a minimum weight of 40 kg. An initial Sentinel Safety Cohort will include 12 healthy volunteers; all other participants in the study will be either immunocompromised or immunocompetent (including healthy participants) with all degrees of SARS-CoV-2 infection risk.
  Interventions: Biological: AZD7442 (EVUSHELD™) (Sub-study) Immunocompromised participants offered AZD3152

INTERVENTIONS:
Biological: AZD5156 (Parent study Sentinel Safety Cohort) — 600 mg AZD5156 consisting of 300 mg AZD1061 at 100 mg/mL and 300 mg AZD3152 at 150 mg/mL
  3 mL of AZD1061 2 mL of AZD3152 IM on Visit 1 Day 1
  Arms: Parent study Sentinel Safety Cohort - Subcohort 1a Gluteal - AZD5156; Parent study Sentinel Safety Cohort - Subcohort 1b Thigh - AZD5156; Parent study Sentinel Safety Cohort - Subcohort 2a Gluteal- AZD5156; Parent study Sentinel Safety Cohort - Subcohort 2b Thigh - AZD5156
Biological: Placebo (Parent study Sentinel Safety Cohort) — single dose of Placebo (3 mL + 2 mL) IM
  Arms: Parent study Main Cohort - AZD3152; Parent study Sentinel Safety Cohort - Subcohort 1a Gluteal - Placebo; Parent study Sentinel Safety Cohort - Subcohort 1b Thigh - Placebo; Parent study Sentinel Safety Cohort - Subcohort 2a Gluteal - Placebo; Parent study Sentinel Safety Cohort - Subcohort 2b Thigh - Placebo
Biological: EVUSHELD™ (Parent study Main Cohort) — 600 mg EVUSHELD™/AZD7442 consisting of 300 mg AZD1061 and 300 mg AZD8895, both at 100 mg/mL
  2 IM injections (thigh) of 3 mL each IM on Visit 1 Day 1 and on Visit 5 Day 181
  Other Names: EVUSHELD™
  Arms: Parent study Main Cohort - EVUSHELD™
Biological: AZD3152 (Parent study Main Cohort) — 300 mg AZD3152 at 150 mg/mL
  1 IM injection (thigh) of 2 mL of AZD3152 on Visit 1 Day 1 and on Visit 5 Day 181
  Arms: Parent study Main Cohort - AZD3152
Biological: Placebo (Parent study Main Cohort) — Single doses of 0.9% sodium chloride 2 mL IM for injection on Visit 1 Day 1 and Visit 5 Day 181
  Arms: Parent study Main Cohort - Placebo
Biological: AZD3152 (Sub-study) — Single dose of 1200 mg IV at Visit 1 Day 1
  Arms: Sub-study - AZD3152
Biological: AZD7442 - EVUSHELD™ (Sub-study) — Single dose 300 mg IM administered on Visit 1 Day 1
  Arms: Sub-study - AZD7442 (EVUSHELD™)
Biological: AZD7442 (EVUSHELD™) (Sub-study) Immunocompromised participants offered AZD3152 — Single dose of AZD7442 (EVUSHELD™) 300 mg IM
  Arms: Sub-study - AZD7442 (EVUSHELD™) Immunocompromised participants offered AZD3152 1200mg IV

SUMMARY:
AZD3152, a single mAb, is being developed to have broad neutralizing activity across known SARS-CoV-2 variants of concern for pre-exposure prophylaxis of COVID-19.

The aim of the Phase I/III study (Parent Study) will be to evaluate the safety, efficacy and neutralizing activity of AZD3152 compared with comparator for pre exposure prophylaxis of COVID-19, and separately evaluate the safety and PK of AZD5156, a combination of AZD3152 and AZD1061.

Sub-study:

This Phase II sub-study of SUPERNOVA will assess the safety, PK, and predicted neutralizing activity of AZD3152 compared with EVUSHELD for pre-exposure prophylaxis of COVID-19.

DETAILED DESCRIPTION:
In the Parent study, the Phase I Sentinel Safety Cohort will assess the safety of AZD5156 (a combination of 2 mAbs, AZD1061 [cilgavimab, a component of AZD7442 (EVUSHELD)] and AZD3152) in healthy adults and the Phase III Main Cohort will assess the safety, efficacy, PK, and neutralizing activity of two doses of AZD3152 compared with two doses of comparator given at a 6-month interval in adults and adolescents 12 years of age or older (weighing at least 40 kg) with conditions causing immune impairment, who are less likely to mount an adequate protective immune response after vaccination and thus are at higher risk of developing severe COVID-19 in 18 countries.

Sub-study:

This Phase II sub-study of SUPERNOVA is operating in USA only, and it will assess the safety, PK, and predicted neutralizing activity of AZD3152 in adults 18 years of age or older (weighing at least 40 kg) with conditions causing immune impairment who are less likely to mount an adequate protective immune response after vaccination as well as individuals who are immunocompetent (including healthy participants) with all degrees of SARS-CoV-2 infection risk.

ELIGIBILITY:
Parent study - Sentinel Safety Cohort Participants (Phase I):

Parent study - Sentinel Cohort Inclusion Criteria:

* Healthy participants according to medical history, physical examination, baseline safety laboratory tests, and screening parameters, according to the judgment of the investigator, with no concomitant disease or concomitant medication (except for medication specifically permitted by the protocol).
* Age 18 to 55 years at the time of signing the informed consent.
* Negative rapid antigen test at Visit 1.
* Weight ≥ 45 kg and ≤ 110 kg at screening.

Parent study - Sentinel Cohort Exclusion Criteria:

* Women who are pregnant, lactating, or of childbearing potential and not using a highly effective method of contraception or abstinence from at least 4 weeks prior to study intervention administration and until at least 6 months after study intervention administration.
* Known hypersensitivity to any component of the study intervention.
* Previous hypersensitivity or severe adverse reaction following administration of a mAb.
* Acute (time-limited) or febrile (temperature ≥ 38.0°C [100.4ºF]) illness/infection on day prior to or day of planned dosing; participants excluded for transient acute illness may be dosed if illness resolves within the screening period or may be rescreened once.
* Blood drawn in excess of a total of 450 mL (1 unit) for any reason within 30 days prior to Visit 1.
* Clinically significant bleeding disorder (eg, factor deficiency, coagulopathy, or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture.
* Receipt of immunoglobulin (non-COVID related) or blood products within 6 months prior to Visit 1.
* Previous receipt of a mAb against SARS-CoV-2.
* Receipt of a COVID-19 vaccine within 3 months prior to Visit 1.
* Receipt of a COVID-19 antiviral for prophylaxis within 3 months prior to Visit 1
* COVID-19 within 3 months prior to Visit 1 (confirmed either by laboratory testing or a rapid test [including at home testing]).
* Receipt of any IMP in the preceding 90 days or expected receipt of IMP during the period of study follow-up, or concurrent participation in another interventional study.
* Known or suspected congenital or acquired immunodeficiency, or receipt of immunosuppressive therapy, including any course of glucocorticoid therapy exceeding 2 weeks of prednisone or equivalent at a dose of 20 mg daily or every other day within 6 months prior to screening.
* Active infection with hepatitis B or C.
* Serum creatinine, AST, or ALT above 1.5 × ULN at screening
* History of malignancy other than treated non-melanoma skin cancers or locally-treated cervical cancer in previous 5 years.

Parent study - Main Cohort Participants (Phase III):

Parent study - Main Cohort Inclusion Criteria:

* Participant must be 12 years of age or older at the time of signing the informed consent.
* Negative rapid antigen test prior to dosing at Visit 1.
* Weight ≥ 40 kg at screening.
* Participants must satisfy at least 1 of the following risk factors at enrollment:

  * Have solid tumor cancer and be on active immunosuppressive treatment
  * Have hematologic malignancy
  * Transplant participants must satisfy at least one of the following:

    1. Have had a solid organ transplant within 2 years and / or
    2. Had a hematopoietic stem cell transplant within 2 years and / or
    3. Who have chronic graft-versus-host disease
    4. Participants who previously had a solid organ transplant or hematopoietic stem cell transplant more than 2 years prior to Visit 1 may also be eligible based on the inclusion criterion for immunosuppressive treatment
  * Are actively taking immunosuppressive medicines (eg, are using corticosteroids [ie, ≥ 20 mg prednisone or equivalent per day when administered for ≥ 2 weeks], high dose alkylating agents, antimetabolites, transplant-related immunosuppressive drugs, cancer chemotherapeutic agents classified as severely immunosuppressive [eg, Bruton's tyrosine kinase inhibitors], tumor-necrosis blockers, or other immunosuppressive or immunomodulatory biologic agents (eg, for rheumatic diseases)
  * Received chimeric antigen receptor T cell therapy
  * Within 1 year of receiving B-cell depleting therapies (eg, rituximab, ocrelizumab, ofatumumab, alemtuzumab)
  * Have a moderate or severe primary (eg, DiGeorge syndrome) or secondary (eg, hemodialysis) immunodeficiency
  * Advanced or untreated HIV infection (people with HIV and CD4 cell counts < 200/mm3 within 6 months of Visit 1, history of an AIDS-defining illness without immune reconstitution, or clinical manifestations of symptomatic HIV)
* Medically stable defined as disease not requiring significant change in maintenance therapy or hospitalization for worsening disease or any recent CV event (eg, acute myocardial infarction, thromboembolic event) during the 1 month prior to enrollment, with no acute change in condition at the time of study enrollment as judged by the Investigator and no expected changes at the time of the enrollment.
* Able to understand and comply with all study requirements/procedures (if applicable, with assistance by caregiver, surrogate, or legally authorized representative or equivalent representative as locally defined), including those at Illness Visits, based on the assessment of the Investigator.

Parent study - Main Cohort Exclusion Criteria:

* Women who are pregnant, lactating, or of childbearing potential and not using a highly effective method of contraception or abstinence from at least 4 weeks prior to study intervention administration and until at least 6 months after study intervention administration. Note: female participants aged > 12 years will be considered to be a woman of childbearing potential.
* Known hypersensitivity to any component of the study intervention.
* Previous hypersensitivity or severe adverse reaction following administration of a mAb.
* Acute (time-limited) or febrile (temperature ≥ 38.0°C [100.4ºF]) illness/infection on day prior to or day of planned dosing; participants excluded for transient acute illness may be dosed if illness resolves and may be rescreened for enrollment once.
* Blood drawn in excess of a total of 450 mL (1 unit) for any reason within 30 days prior to Visit 1.
* Clinically significant bleeding disorder (eg, factor deficiency, coagulopathy, or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture.
* Receipt of IV or SC immunoglobulin within 6 months prior to Visit 1 or expected to receive IV or SC immunoglobulin 6 months after dosing.
* Receipt of convalescent COVID-19 plasma treatment within 6 months prior to Visit 1.
* Previous receipt of a mAb against SARS-CoV-2 within 6 months prior to Visit 1.
* Receipt of a COVID-19 vaccine within 3 months prior to Visit 1.
* Receipt of a COVID-19 antiviral for prophylaxis within at least 2 weeks prior to Visit 1.
* COVID-19 within 3 months prior to Visit 1 (confirmed either by laboratory testing or a rapid test [including at home testing]).
* Receipt of any IMP in the preceding 90 days or expected receipt of IMP during the period of study follow-up, or concurrent participation in another interventional study except where the participant ceased IMP treatment >90 days and is in the follow-up period of the study and not expected to receive further IMP).

Sub-study - Inclusion Criteria (Phase II):

Sub-study - Sentinel Safety Cohort Inclusion Criteria:

* Healthy, defined according to medical history, physical examination, baseline safety laboratory tests, and screening parameters, according to the judgment of the Investigator.
* Participants must be 18 to 55 years at the time of signing the informed consent.
* Weight ≥ 45 kg and ≤ 110 kg at screening.

Sub-study - Full Sub-study Cohort Inclusion Criteria:

* Immunocompromised or immunocompetent, including healthy participants, with all degrees of SARS-CoV-2 infection risk, will be enrolled following completion of Sentinel Safety Cohort enrolment.
* Participants must be 18 years of age or older at the time of signing the informed consent.
* Weight ≥ 40 kg at screening.

Sub-study - Sub-study Sentinel Safety Cohort and Full Sub-study Cohort Inclusion Criteria:

* Written informed consent and any locally required authorization (eg, HIPAA in the US) obtained from the participant prior to performing any protocol-related procedures, including screening evaluations.
* Negative rapid antigen test for SARS-CoV-2 prior to dosing at Visit 1.
* Medically stable defined as disease not requiring significant change in maintenance therapy or hospitalization for worsening disease or any recent cardiovascular event (eg, acute myocardial infarction, thromboembolic event) during the 1 month prior to enrollment, with no acute change in condition at the time of study enrollment as judged by the Investigator and no expected changes at the time of the enrollment.
* Able to understand and comply with all study requirements/procedures (if applicable, with assistance by caregiver, surrogate, or legally authorized representative or equivalent representative as locally defined), based on the assessment of the Investigator.

Sub-study - Exclusion Criteria (Phase II):

Sub-study - Sentinel Safety Cohort Exclusion Criteria:

* Active infection with hepatitis B or C.
* Serum creatinine, AST, or ALT above 1.5 × ULN at screening.
* History of malignancy other than treated non-melanoma skin cancers or locally-treated cervical cancer in previous 5 years.

Sub-study - Sentinel Safety Cohort and Full Sub-study Cohort Exclusion Criteria:

* Receipt of EVUSHELD (AZD7442) within 12 months prior to Visit 1.
* Women who are pregnant, lactating, or of childbearing potential and not using a highly effective method of contraception or abstinence from at least 4 weeks prior to study intervention administration and until at least 6 months after study intervention administration. Note: female participants aged > 12 years will be considered to be a woman of childbearing potential.
* Known hypersensitivity to any component of the study intervention.
* Previous hypersensitivity or severe adverse reaction following administration of a mAb.
* Acute (time-limited) or febrile (temperature ≥ 38.0°C [100.4ºF]) illness/infection on day prior to or day of planned dosing; participants excluded for transient acute illness may be dosed if illness resolves and may be rescreened for enrollment once.
* Blood drawn in excess of a total of 450 mL (1 unit) for any reason within 30 days prior to Visit 1.
* Clinically significant bleeding disorder (eg, factor deficiency, coagulopathy, or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture.
* Has human immunodeficiency virus infection.
* Receipt of IV or SC immunoglobulin or blood products within 6 months prior to Visit 1 and expected to receive IV or SC immunoglobulin or blood products 6 months after dosing.
* Receipt of a COVID-19 vaccine within 3 months prior to Visit 1.
* Receipt of a COVID-19 antiviral for prophylaxis within at least 2 weeks prior to Visit 1.
* COVID-19 within 3 months prior to Visit 1 (confirmed either by laboratory RT-PCR testing or a rapid antigen test [including at-home testing]).
* Receipt of any IMP in the preceding 90 days or expected receipt of IMP during the period of study follow-up, or concurrent participation in another interventional study (except where the participant ceased IMP treatment > 90 days and is in the follow-up period of the study and not expected to receive further IMP).

Ages: 12 Years to 130 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3882 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Parent study - Sentinel Safety Cohort: To evaluate the safety of AZD5156 | AEs will be collected from IMP administration approximately 90 days following. AESIs will be collected from IMP administration through to Visit 11 (Day 361). SAEs and MAAEs will be collected up to Visit 11 (Day 361).
  Occurence of AEs, SAEs, MAAEs, and AESIs will be collected throughout the study
Parent study - Main Cohort: To evaluate the safety of AZD3152 and EVUSHELD and/or placebo | Occurrence of AEs collected through approximately 90 days after each IMP administration through to Visit 10 (Day 451). SAEs and MAAEs will be collected up to Visit 10 (Day 451).
  Occurrence of AEs, SAEs, MAAEs, and AESIs will be collected throughout the study
Parent study-Main cohort: To compare the efficacy of AZD3152 to EVUSHELD and/or placebo in the prevention of symptomatic COVID 19 caused by any SARS-CoV-2 variant | Confirmed symptomatic COVID-19 case is evaluated from first dose up to 181 days after last dose. For participants that receive two doses, the evaluation period would be approximately 361 days.
  Endpoint: Confirmed symptomatic COVID-19 case, classified as a binary outcome incorporating the time from the first dose of IMP until a participant develops their first symptoms for COVID-19 or are censored. Summary measure: Prophylactic efficacy, calculated as 1 - Hazard Ratio (HR) (AZD3152 versus EVUSHELD and/or placebo) using a hazard regression model.
Parent study - Main cohort: To compare the efficacy of AZD3152 to EVUSHELD and/or placebo in the prevention of symptomatic COVID 19 attributable to matched variants (variants that do not contain the F456L mutation) | Confirmed symptomatic COVID-19 case is evaluated from first dose up to 181 days after last dose. For participants that receive two doses, the evaluation period would be approximately 361 days.
  Endpoint: Confirmed symptomatic COVID-19 case attributable to matched variants, classified as a binary outcome incorporating the time from the first dose of IMP until a participant develops their first symptoms for COVID-19 or are censored. Summary measure: Prophylactic efficacy, calculated as 1 - Hazard Ratio (HR) (AZD3152 versus EVUSHELD and/or placebo) using a hazard regression model.
Sub-study: To evaluate the safety of AZD3152 and EVUSHELD | SAEs, MAAEs, and AESIs collected throughout the study for the final analysis.
  Occurrence of AEs collected through 29 days after IMP administration for the primary analysis.
Sub-study: To compare the SARS-CoV-2 nAb responses to a current VOC following AZD3152 administration vs SARS-CoV-2 nAb responses to prior variants following EVUSHELD administration | Predicted GMT ratio of SARS-CoV-2 nAbs between the treatment arms at Visit 3 (Day 29) for the variant that each IMP is intended to neutralize.
  SARS-CoV-2 nAb responses to a current VOC following AZD3152 administration vs SARS-CoV-2 nAb responses to prior variants following EVUSHELD administration.

SECONDARY OUTCOMES:
Parent study - Sentinel Safety Cohort: To characterize the Pharmacokinetics of AZD5156 (AZD1061 and AZD3152) in serum. | Samples will be collected from Visit 1 (Day 1) up to Visit 11 (Day 361).
  AZD5156 (AZD1061 and AZD3152) serum concentrations at each visit.
Parent study - Sentinel Safety Cohort: To characterize the Pharmacokinetics parameter of maximum concentration (Cmax) of AZD5156 (AZD1061 and AZD3152) in serum | Samples will be collected from Visit 1 (Day 1) up to Visit 11 (Day 361)
  To describe maximum concentration (Cmax) for AZD5156 (AZD1061 and AZD3152).
Parent study - Sentinel Safety Cohort: To characterize the Pharmacokinetics parameter of time to maximum serum concentration (tmax) of AZD5156 (AZD1061 and AZD3152) in serum | Samples will be collected from Visit 1 (Day 1) up to Visit 11 (Day 361).
  To describe time to maximum serum concentration (tmax) for AZD5156 (AZD1061 and AZD3152).
Parent study - Sentinel Safety Cohort: To characterize the Pharmacokinetics parameter of terminal half-life (t½) of AZD5156 (AZD1061 and AZD3152) in serum | Samples will be collected from Visit 1 (Day 1) up to Visit 11 (Day 361).
  To describe terminal half-life (t½) for AZD5156 (AZD1061 and AZD3152).
Parent study - Sentinel Safety Cohort: To characterize the Pharmacokinetics parameter of area under the concentration-time curve at the last measured time point (AUClast) of AZD5156 (AZD1061 and AZD3152) in serum | Samples will be collected from Visit 1 (Day 1) up to Visit 11 (Day 361).
  To describe area under the concentration-time curve at the last measured time point (AUClast) for AZD5156 (AZD1061 and AZD3152).
Parent study - Sentinel Safety Cohort: To characterize the Pharmacokinetics parameter of area under the concentration-time curve from time zero extrapolated to infinity (AUCinf) of AZD5156 (AZD1061 and AZD3152) in serum | Samples will be collected from visit 1 (Day 1) up to visit 11 (Day 361).
  To describe area under the concentration-time curve from time zero extrapolated to infinity (AUCinf) for AZD5156 (AZD1061 and AZD3152).
Parent study - Sentinel Safety Cohort: To evaluate the ADA responses to AZD5156, AZD3152, and AZD1061 in serum | Samples will be collected from Visit 1 (Day 1) up to Visit 11 (Day 361)
  Incidence of ADA to AZD5156, AZD3152, and AZD1061, ADA titers
Parent study - Main Cohort: To compare the nAb responses to the SARS-CoV-2 variants Alpha, Omicron BA.2, Omicron BA.4/5 and/or Omicron XBB.1.5 in serum following AZD3152 and EVUSHELD and/or placebo administration | Visit 3 (Day 29)
  GMT and GMFR ratio of SARS-CoV-2 nAbs between the treatment arms at Visit 3 (Day 29).
  Descriptive statistics for GMTs and GMFRs will be provided.
Parent study - Main Cohort: To describe the incidence of symptomatic COVID-19, severe COVID-19, COVID-19 related hospitalization, and COVID-19 related death in participants receiving study intervention | COVID-19 incidence variables to be evaluated through Visit 9 (Day 361)
  Incidence of a post-treatment:
  * Symptomatic COVID-19 case (negative RT-PCR at baseline to positive at any time up to 6 and 12 months) caused by any SARS-CoV-2 variant
  * Symptomatic COVID-19 case (negative RT-PCR at baseline to positive at any time up to 6 and 12 months) caused by any SARS-CoV-2 matched variants
  * Severe COVID-19 caused by any SARS-CoV-2 variant
  * Severe COVID-19 caused by any SARS-CoV-2 matched variants
  * Composite of COVID-19 related hospitalization and/or COVID-19 related death (WHO COVID-19 Clinical Progression Scale score ≥ 4)
  * COVID-19 related hospitalization (separately)
  * COVID-19 related death (separately)
Parent study - Main Cohort: To characterize the Pharmacokinetics (PK)of the AZD3152 and AZD7442 (AZD1061 and AZD8865) in serum concentrations at each visit. | Samples will be collected from Visit 1 (Day 1) up to Visit 9 (Day 361)
  AZD3152 and AZD7442 (AZD1061 and AZD8895) serum concentrations at each visit.
Parent study - Main Cohort: To evaluate the Anti-drug Antibodies (ADA) responses to AZD3152 and AZD7442 in serum | Samples will be collected from Visit 1 (Day 1) up to Visit 9 (Day 361)
  Incidence of Anti-drug Antibodies (ADA) to AZD3152, AZD7442, AZD1061, and AZD8895, ADA titers
Sub-study: To characterize the Pharmacokinetics of AZD3152 and AZD7442 (EVUSHELD) in serum | Samples will be collected from Visit 1 (Day 1) up to Visit 5 (Day 181).
  AZD3152, AZD7442 (EVUSHELD), cilgavimab, and tixagevimab concentrations in serum, over time
Sub-study:To evaluate the ADA response to AZD3152 and AZD7442 (EVUSHELD) in serum | Samples will be collected from Visit 1 (Day 1) up to Visit 5 (Day 181).
  Incidence of ADA to AZD3152, AZD7442 (EVUSHELD), cilgavimab, and tixagevimab; ADA titers

CONTACTS AND LOCATIONS:
Locations (180):
- United States (111):
  - Research Site, Birmingham, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Glendale, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Colton, California
  - Research Site, La Mesa, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Modesto, California
  - Research Site, Sacramento, California
  - Research Site, Tustin, California
  - Research Site, Westminster, California
  - Research Site, Aurora, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Fort Collins, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Coral Gables, Florida
  - Research Site, Fleming Island, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Lake Worth, Florida
  - Research Site, Largo, Florida
  - Research Site, Lauderdale Lakes, Florida
  - Research Site, Leesburg, Florida
  - Research Site, Medley, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Miami Springs, Florida
  - Research Site, North Miami Beach, Florida
  - Research Site, Orlando, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Port Orange, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Burr Ridge, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Gurnee, Illinois
  - Research Site, Evansville, Indiana
  - Research Site, South Bend, Indiana
  - Research Site, West Des Moines, Iowa
  - Research Site, Overland Park, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Bowling Green, Kentucky
  - Research Site, Lexington, Kentucky
  - Research Site, Lake Charles, Louisiana
  - Research Site, Metairie, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Methuen, Massachusetts
  - Research Site, Springfield, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Farmington Hills, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Novi, Michigan
  - Research Site, Saint Clair Shores, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Jefferson City, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Missoula, Montana
  - Research Site, Lincoln, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Portsmouth, New Hampshire
  - Research Site, Hackensack, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Buffalo, New York
  - Research Site, Ridgewood, New York
  - Research Site, Rochester, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Monroe, North Carolina
  - Research Site, Morehead City, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Westlake, Ohio
  - Research Site, Allentown, Pennsylvania
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Harrisburg, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, North Charleston, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Knoxville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, Kingwood, Texas
  - Research Site, Mesquite, Texas
  - Research Site, San Angelo, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Shenandoah, Texas
  - Research Site, Layton, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Annandale, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Olympia, Washington
  - Research Site, Seattle, Washington
  - Research Site, Madison, Wisconsin
- Australia (6):
  - Research Site, Melbourne
  - Research Site, Murdoch
  - Research Site, Parkville
  - Research Site, Raymond Terrace
  - Research Site, Sippy Downs
  - Research Site, West Perth
- Belgium (2):
  - Research Site, Alken
  - Research Site, Liège
- Research Site, Montreal, Quebec, Canada
- Denmark (5):
  - Research Site, Aalborg
  - Research Site, Aarhus
  - Research Site, Hvidovre
  - Research Site, Roskilde
  - Research Site, Svendborg
- France (11):
  - Research Site, Dijon
  - Research Site, La Roche-sur-Yon
  - Research Site, Lille
  - Research Site, Nantes
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Poitiers
  - Research Site, Saint-Etienne
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Tours
- Germany (5):
  - Research Site, Cologne
  - Research Site, Essen
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Mainz
- Israel (2):
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
- Malaysia (4):
  - Research Site, Kuala Lumpur
  - Research Site, Kuching
  - Research Site, Seberang Jaya
  - Research Site, Sunway City
- Poland (2):
  - Research Site, Krakow
  - Research Site, Skórzewo
- Research Site, Singapore, Singapore
- South Korea (2):
  - Research Site, Gyeonggi-do
  - Research Site, Seoul
- Spain (9):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Madrid
  - Research Site, Marbella (Málaga)
  - Research Site, Mérida
  - Research Site, Pozuelo de Alarcón
  - Research Site, Valladolid
  - Research Site, Vigo
- Taiwan (2):
  - Research Site, Taichung
  - Research Site, Taipei
- Thailand (3):
  - Research Site, Bangkok
  - Research Site, Khon Kaen
  - Research Site, Muang
- Research Site, Abu Dhabi, United Arab Emirates
- United Kingdom (11):
  - Research Site, Bristol
  - Research Site, Edinburgh
  - Research Site, Harrow
  - Research Site, Leeds
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Oxford
  - Research Site, Sheffield
  - Research Site, Torpoint
  - Research Site, Truro
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Hochiminh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Background] Alhumaid S, Al Mutair A, Al Alawi Z, Rabaan AA, Tirupathi R, Alomari MA, Alshakhes AS, Alshawi AM, Ahmed GY, Almusabeh HM, Alghareeb TT, Alghuwainem AA, Alsulaiman ZA, Alabdulmuhsin MA, AlBuwaidi EA, Dukhi AKB, Mufti HN, Al-Qahtani M, Dhama K, Al-Tawfiq JA, Al-Omari A. Anaphylactic and nonanaphylactic reactions to SARS-CoV-2 vaccines: a systematic review and meta-analysis. Allergy Asthma Clin Immunol. 2021 Oct 16;17(1):109. doi: 10.1186/s13223-021-00613-7. PMID 34656181
- [Background] Bosch BJ, van der Zee R, de Haan CA, Rottier PJ. The coronavirus spike protein is a class I virus fusion protein: structural and functional characterization of the fusion core complex. J Virol. 2003 Aug;77(16):8801-11. doi: 10.1128/jvi.77.16.8801-8811.2003. PMID 12885899
- [Background] CDC 2021 CDC (Centers for Disease Control and Prevention). General Best Practice Guidelines for Immunization: Altered Immunocompetence. Available from: https://www.cdc.gov/vaccines/hcp/acip-recs/general-recs/immunocompetence.html. Accessed 23 May 2022.
- [Background] Case JB, Mackin S, Errico JM, Chong Z, Madden EA, Whitener B, Guarino B, Schmid MA, Rosenthal K, Ren K, Dang HV, Snell G, Jung A, Droit L, Handley SA, Halfmann PJ, Kawaoka Y, Crowe JE Jr, Fremont DH, Virgin HW, Loo YM, Esser MT, Purcell LA, Corti D, Diamond MS. Resilience of S309 and AZD7442 monoclonal antibody treatments against infection by SARS-CoV-2 Omicron lineage strains. Nat Commun. 2022 Jul 2;13(1):3824. doi: 10.1038/s41467-022-31615-7. PMID 35780162
- [Background] Dall'Acqua WF, Kiener PA, Wu H. Properties of human IgG1s engineered for enhanced binding to the neonatal Fc receptor (FcRn). J Biol Chem. 2006 Aug 18;281(33):23514-24. doi: 10.1074/jbc.M604292200. Epub 2006 Jun 21. PMID 16793771
- [Background] Fact Sheet EUA Bebtelovimab 2022 US Food and Drug Administration. Fact Sheet For Healthcare Providers: Emergency Use Authorization for Bebtelovimab, March 2022. Available at: https://www.fda.gov/media/156152/download. Accessed 23 May 2022.
- [Background] Gupta A, Gonzalez-Rojas Y, Juarez E, Crespo Casal M, Moya J, Falci DR, Sarkis E, Solis J, Zheng H, Scott N, Cathcart AL, Hebner CM, Sager J, Mogalian E, Tipple C, Peppercorn A, Alexander E, Pang PS, Free A, Brinson C, Aldinger M, Shapiro AE; COMET-ICE Investigators. Early Treatment for Covid-19 with SARS-CoV-2 Neutralizing Antibody Sotrovimab. N Engl J Med. 2021 Nov 18;385(21):1941-1950. doi: 10.1056/NEJMoa2107934. Epub 2021 Oct 27. PMID 34706189
- [Background] Harpaz R, Dahl RM, Dooling KL. Prevalence of Immunosuppression Among US Adults, 2013. JAMA. 2016 Dec 20;316(23):2547-2548. doi: 10.1001/jama.2016.16477. No abstract available. PMID 27792809
- [Background] Hoffmann M, Kleine-Weber H, Schroeder S, Kruger N, Herrler T, Erichsen S, Schiergens TS, Herrler G, Wu NH, Nitsche A, Muller MA, Drosten C, Pohlmann S. SARS-CoV-2 Cell Entry Depends on ACE2 and TMPRSS2 and Is Blocked by a Clinically Proven Protease Inhibitor. Cell. 2020 Apr 16;181(2):271-280.e8. doi: 10.1016/j.cell.2020.02.052. Epub 2020 Mar 5. PMID 32142651
- [Background] Levin MJ, Ustianowski A, De Wit S, Launay O, Avila M, Templeton A, Yuan Y, Seegobin S, Ellery A, Levinson DJ, Ambery P, Arends RH, Beavon R, Dey K, Garbes P, Kelly EJ, Koh GCKW, Near KA, Padilla KW, Psachoulia K, Sharbaugh A, Streicher K, Pangalos MN, Esser MT; PROVENT Study Group. Intramuscular AZD7442 (Tixagevimab-Cilgavimab) for Prevention of Covid-19. N Engl J Med. 2022 Jun 9;386(23):2188-2200. doi: 10.1056/NEJMoa2116620. Epub 2022 Apr 20. PMID 35443106
- [Background] Li F. Structure, Function, and Evolution of Coronavirus Spike Proteins. Annu Rev Virol. 2016 Sep 29;3(1):237-261. doi: 10.1146/annurev-virology-110615-042301. Epub 2016 Aug 25. PMID 27578435
- [Background] Loo YM, McTamney PM, Arends RH, Abram ME, Aksyuk AA, Diallo S, Flores DJ, Kelly EJ, Ren K, Roque R, Rosenthal K, Streicher K, Tuffy KM, Bond NJ, Cornwell O, Bouquet J, Cheng LI, Dunyak J, Huang Y, Rosenbaum AI, Pilla Reddy V, Andersen H, Carnahan RH, Crowe JE Jr, Kuehne AI, Herbert AS, Dye JM, Bright H, Kallewaard NL, Pangalos MN, Esser MT. The SARS-CoV-2 monoclonal antibody combination, AZD7442, is protective in nonhuman primates and has an extended half-life in humans. Sci Transl Med. 2022 Mar 9;14(635):eabl8124. doi: 10.1126/scitranslmed.abl8124. Epub 2022 Mar 9. PMID 35076282
- [Background] Lusvarghi S, Pollett SD, Neerukonda SN, Wang W, Wang R, Vassell R, Epsi NJ, Fries AC, Agan BK, Lindholm DA, Colombo CJ, Mody R, Ewers EC, Lalani T, Ganesan A, Goguet E, Hollis-Perry M, Coggins SA, Simons MP, Katzelnick LC, Wang G, Tribble DR, Bentley L, Eakin AE, Broder CC, Erlandson KJ, Laing ED, Burgess TH, Mitre E, Weiss CD. SARS-CoV-2 BA.1 variant is neutralized by vaccine booster-elicited serum but evades most convalescent serum and therapeutic antibodies. Sci Transl Med. 2022 May 18;14(645):eabn8543. doi: 10.1126/scitranslmed.abn8543. Epub 2022 May 18. PMID 35380448
- [Background] Maltezou HC, Anastassopoulou C, Hatziantoniou S, Poland GA, Tsakris A. Anaphylaxis rates associated with COVID-19 vaccines are comparable to those of other vaccines. Vaccine. 2022 Jan 21;40(2):183-186. doi: 10.1016/j.vaccine.2021.11.066. Epub 2021 Nov 27. PMID 34863620
- [Background] NIH 2017 NIH. Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. Available at: https://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm#ctc_50. Published 2017. Accessed 23 May 2022.
- [Background] Oganesyan V, Gao C, Shirinian L, Wu H, Dall'Acqua WF. Structural characterization of a human Fc fragment engineered for lack of effector functions. Acta Crystallogr D Biol Crystallogr. 2008 Jun;64(Pt 6):700-4. doi: 10.1107/S0907444908007877. Epub 2008 May 14. PMID 18560159
- [Background] Parker EPK, Desai S, Marti M, Nohynek H, Kaslow DC, Kochhar S, O'Brien KL, Hombach J, Wilder-Smith A. Response to additional COVID-19 vaccine doses in people who are immunocompromised: a rapid review. Lancet Glob Health. 2022 Mar;10(3):e326-e328. doi: 10.1016/S2214-109X(21)00593-3. No abstract available. PMID 35180408
- [Background] Sampson HA, Munoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, Brown SG, Camargo CA Jr, Cydulka R, Galli SJ, Gidudu J, Gruchalla RS, Harlor AD Jr, Hepner DL, Lewis LM, Lieberman PL, Metcalfe DD, O'Connor R, Muraro A, Rudman A, Schmitt C, Scherrer D, Simons FE, Thomas S, Wood JP, Decker WW. Second symposium on the definition and management of anaphylaxis: summary report--Second National Institute of Allergy and Infectious Disease/Food Allergy and Anaphylaxis Network symposium. J Allergy Clin Immunol. 2006 Feb;117(2):391-7. doi: 10.1016/j.jaci.2005.12.1303. PMID 16461139
- [Background] Tuekprakhon A, Nutalai R, Dijokaite-Guraliuc A, Zhou D, Ginn HM, Selvaraj M, Liu C, Mentzer AJ, Supasa P, Duyvesteyn HME, Das R, Skelly D, Ritter TG, Amini A, Bibi S, Adele S, Johnson SA, Constantinides B, Webster H, Temperton N, Klenerman P, Barnes E, Dunachie SJ, Crook D, Pollard AJ, Lambe T, Goulder P, Paterson NG, Williams MA, Hall DR; OPTIC Consortium; ISARIC4C Consortium; Fry EE, Huo J, Mongkolsapaya J, Ren J, Stuart DI, Screaton GR. Antibody escape of SARS-CoV-2 Omicron BA.4 and BA.5 from vaccine and BA.1 serum. Cell. 2022 Jul 7;185(14):2422-2433.e13. doi: 10.1016/j.cell.2022.06.005. Epub 2022 Jun 9. PMID 35772405
- [Background] Walls AC, Tortorici MA, Snijder J, Xiong X, Bosch BJ, Rey FA, Veesler D. Tectonic conformational changes of a coronavirus spike glycoprotein promote membrane fusion. Proc Natl Acad Sci U S A. 2017 Oct 17;114(42):11157-11162. doi: 10.1073/pnas.1708727114. Epub 2017 Oct 3. PMID 29073020
- [Background] Weinreich DM, Sivapalasingam S, Norton T, Ali S, Gao H, Bhore R, Musser BJ, Soo Y, Rofail D, Im J, Perry C, Pan C, Hosain R, Mahmood A, Davis JD, Turner KC, Hooper AT, Hamilton JD, Baum A, Kyratsous CA, Kim Y, Cook A, Kampman W, Kohli A, Sachdeva Y, Graber X, Kowal B, DiCioccio T, Stahl N, Lipsich L, Braunstein N, Herman G, Yancopoulos GD; Trial Investigators. REGN-COV2, a Neutralizing Antibody Cocktail, in Outpatients with Covid-19. N Engl J Med. 2021 Jan 21;384(3):238-251. doi: 10.1056/NEJMoa2035002. Epub 2020 Dec 17. PMID 33332778
- [Background] WHO 2022 World Health Organization. WHO COVID-19 Case definition, July 2022. Available at: https://www.who.int/publications/i/item/WHO-2019-nCoV-Surveillance_Case_Definition 2022.1. Accessed 05 May 2023.
- [Background] WHO 2023 WHO Coronavirus disease (COVID-19) dashboard. Available at: https://covid19.who.int. Accessed 05 June 2023.
- [Background] Kelly JD, Leonard S, Hoggatt KJ, Boscardin WJ, Lum EN, Moss-Vazquez TA, Andino R, Wong JK, Byers A, Bravata DM, Tien PC, Keyhani S. Incidence of Severe COVID-19 Illness Following Vaccination and Booster With BNT162b2, mRNA-1273, and Ad26.COV2.S Vaccines. JAMA. 2022 Oct 11;328(14):1427-1437. doi: 10.1001/jama.2022.17985. PMID 36156706
- [Derived] Haidar G, Thomas S, Loubet P, Baker RI, Benfield T, Boonyaratanakornkit J, Kiertiburanakul S, Kim AHJ, Longbrake EE, Molina JM, Paredes R, Tucker D, Uriel A, Weinmann-Menke J, Aksyuk AA, Clegg LE, Currie A, Yang H, Flyrin K, Gibbs M, Shroff M, Perez JL, Chang LJ, Cohen TS; SUPERNOVA study group. Efficacy and safety of sipavibart for prevention of COVID-19 in individuals who are immunocompromised (SUPERNOVA): a randomised, controlled, double-blind, phase 3 trial. Lancet Infect Dis. 2025 Jul;25(7):813-826. doi: 10.1016/S1473-3099(24)00804-1. Epub 2025 Feb 24. PMID 40015292
- [Derived] Cai Y, Diallo S, Rosenthal K, Ren K, Flores DJ, Dippel A, Oganesyan V, van Dyk N, Chen X, Cantu E, Choudhary R, Sulikowski M, Adissu H, Chawla B, Kar S, Liu C, Dijokaite-Guraliuc A, Mongkolsapaya J, Rajan S, Loo YM, Beavon R, Webber C, Chang LJ, Thomas S, Clegg L, Zhang H, Screaton GR, Philbin N, Harre M, Selim A, Martinez-Alier N, Uriel A, Cohen TS, Perez JL, Esser MT, Blair W, Francica JR. AZD3152 neutralizes SARS-CoV-2 historical and contemporary variants and is protective in hamsters and well tolerated in adults. Sci Transl Med. 2024 Jun 26;16(753):eado2817. doi: 10.1126/scitranslmed.ado2817. Epub 2024 Jun 26. PMID 38924429